CLINICAL TRIAL: NCT02433509
Title: Phase I Clinical Safety Study About Human Umbilical Cord Blood Monocyte in the Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Buddhist Tzu Chi General Hospital (Other); StemCyte Taiwan Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shinn-Zong Lin, Hualien Tzu Chi Medical Center, Buddhist Tzu Chi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH101-IRB1-114
Record Dates: First submitted 2015-04-21; First posted 2015-05-05 (Estimated); Last update posted 2025-08-06 (Actual); Status verified 2021-11

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; umbilical cord blood
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: acute ischemic stroke
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hUCB w/ Mannitol in acute ischemic stroke (Experimental): 1. The cord blood need to be infusion within less than 10 days after the onset of stroke, with the cord blood mononuclear cells 200 million ~ 500 million will used.
  2. 20% mannitol 200 ml iv for 30±10 min/q8h±2h will be administered twice after cord blood infusion .
  Interventions: Other: hUCB

INTERVENTIONS:
Other: hUCB — 1. The cord blood need to be infusion within less than 10 days after the onset of stroke, and the cord blood mononuclear cells 200 million ~ 500 million will used.
  2. 20% mannitol 200 ml iv for 30±10 min/q8h±2h will be administered twice after cord blood infusion .
  Other Names: 20% Mannnitol

SUMMARY:
The objective of the study is to determine the safely of Human Umbilical Cord Blood mononuclear cells by Intravenous injection in acute ischemic stroke patients.

DETAILED DESCRIPTION:
The study will use Umbilical Cord Blood cells (a special kind of cell that is believed to be a stem cell) isolated from UCB (blood obtained at birth from the umbilical cord blood of babies). StemCyte, a leading accredited UCB banking company with branches in the United States and Taiwan, will provide the units of UCB that match at least 4 out of 6 HLA (human leukocyte antigens) for transplantation. The HLA-matching is the same as that used to match cells and organs for transplantation so that the body does not reject the cells. Then cells injection by Intravenous in acute ischemic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

1. The age of Subjects between 45 through 80 years.
2. Acute Ischemic Stroke.
3. National Institutes of Health Stroke Scale (NIHSS):6-18
4. Brain MRI shows the middle cerebral artery region (M1 and M2) of cerebral i infarction stroke patients.
5. Subjects have no midline shift or hemorrhagic transformation

Exclusion Criteria:

1. NIHSS score reduced more than 4 within after 24 hours.
2. Female are pregnant or lactating.
3. Subjects with impaired liver function, AIDS, cancer or other significant medical condition (including certifiable diseases, rare disease)
4. Subjects joined other clinical trails or received rt-PA therapy.
5. Immune dysfunction or receiving other immunosuppressive agents.
6. Subjects cannot have MRI test
7. Subjects' HLA typing results match less than 4 out of the 6 genotypes

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-05; Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-14 (Actual)

PRIMARY OUTCOMES:
adverse events (AE)and serious adverse reaction(SAE) | after infusion 24, 48, 72 hours , 1 week or discharge , and 1, 3, 6 , 9, 12 months.
  any AE or SAE (related or non-related) during the 12-month follow-up period

SECONDARY OUTCOMES:
Brain Image(MRI) | baseline, after infusion 24 hours, 1, 6, 12months
  changes of Brain Images
abdominal sonography-spleen | baseline, after infusion 24, 72 hours, 3, 12months
  size changes of spleen
NIHSS | baseline, after infusion 24, 48, 72 hours, 1weeks or discharge, 1 3, 6, 9, 12months
  neurology functions change
Berg Balance score | baseline, after infusion 24, 48, 72 hours, 1weeks or discharge, 1 3, 6, 9, 12months
  motor function changes
Barthel Index | baseline, after infusion 24, 48, 72 hours, 1weeks or discharge, 1 3, 6, 9, 12months
  neurology function changes
Blood examination | baseline, after infusion 24, 48, 72 hours, 1 3, 6, 9, 12months
  physical condition monitoring
cytokine family | baseline, after infusion 24, 48, 72 hours, 1 3, 6, 9, 12months
  for study

CONTACTS AND LOCATIONS:
Overall Officials: Shinn-Zong Lin, M.D.;PhD., Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Hualien Tzu Chi Hospital, Hualien City, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No